CLINICAL TRIAL: NCT03558932
Title: IP3R Modulation by Cancer Genes Bcl-2 & PKM2 in Mesothelioma
Brief Title: IP3R Modulation by Cancer Genes in Mesothelioma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Yserbyt Jonas, Principal Investigator, KU Leuven
Other Study IDs: IP3mesov1
Record Dates: First submitted 2018-05-23; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Malignant Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — pleural biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: pleural biopsy — diagnostic sampling

SUMMARY:
Obtaining pleural biopsies in cases of malignant mesothelioma to detect molecular mechnisms and signal transduction

ELIGIBILITY:
Inclusion Criteria:

* suspicion of mesothelioma
* referral for diagnostic thoracoscopy

Exclusion Criteria:

* contra-indication for thoracoscopy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mesothelioma
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Pleural biopsy | 5 years
  Biopsy

OTHER OUTCOMES:
Immunoblotting | 5 years
  biopsy
Cytometric analysis (FACS-based approaches) | 5 years
  biopsy
Live cell imaging for Ca2+-signaling | 5 years
  biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Yserbyt, Principal Investigator — Catholic university Leuven

IPD SHARING:
Plan to Share IPD: No